CLINICAL TRIAL: NCT05954403
Title: National Cohort on Congenital Defects of the Eye: Natural History, Genetic Determinisms and Improved Ocular and Extra-ocular Outcome Prediction for Better Patient Management
Brief Title: National Cohort on Congenital Defects of the Eye
Acronym: RaDiCoACOEIL
Status: Recruiting | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: C15-47
Record Dates: First submitted 2021-12-20; First posted 2023-07-20 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Anophthalmia; Microphthalmia; Aniridia; Anterior Segment Dysgenesis 6, Peters Anomaly Subtype; Anterior Segment Dysgenesis 3, Rieger Subtype
Keywords: Anophthalmia-Microphthalmia-Aniridia; anterior segment dysgenesis; Peters anomaly; Axenfeld-Rieger anomaly; Congenital malformations of the eye; Neuropsychological evaluation
MeSH Terms: conditions — Anophthalmos; Microphthalmos; Aniridia; Iris hypoplasia and glaucoma; Anterior segment mesenchymal dysgenesis; Peters anomaly; Axenfeld-Rieger syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Most of the affected patients have genetic screening of genes involved in ocular developmental defects for diagnosis purpose. Thanks to the organisation of the French geneticists' network, molecular diagnostics of the main genes involved in these ocular defects is centralized in the two principal investigators' laboratory. A panel of 25 genes will be screened by highthroughput sequencing in the laboratory in incident patients and prevalent ones with no previously identified mutation. If no known mutation is identified in a given patient, screening for new genes, once identified as involved in these malformations, will be performed using samples collected and stored at the CHU de Toulouse as part of the current procedure for diagnostic analyses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Congenital malformations of the eye comprise various developmental defects including microphthalmia, anophthalmia, aniridia, and anterior segment anomalies (such as Peters and Axenfeld-Rieger anomalies). These malformations are frequently associated with extra-ocular features and intellectual disability. However, little is known about visual outcome, frequency and consequences of extra-ocular features in patients.

The originality of the project will be to include a spectrum of malformation thought to be a phenotypic continuum (anophthalmia, microphthalmia, aniridia, anterior segment dysgnesis). In addition, we aim to conduct a 10 year follow-up of these children, thus allowing determining ocular and neurological outcomes as any other medical event. We should also be able to determine phenotypic factors that would be associated with good or poor visual and neurologic outcomes

DETAILED DESCRIPTION:
Congenital malformations of the eye include several developmental abnormalities including microphtalmia, aniridia, and anterior segment abnormalities. Microphtalmia is a malformation of the eye that manifests as an eye smaller than normal. In the total absence of visible eyeball is called anophthalmitis. Malformation may concern one or both eyes. Aniridia is characterized by a partial or total absence of the iris. Anterior segment abnormalities include a broad spectrum of malformations affecting the cornea and iris. These are essentially the syndromes of Peters, Rieger and Axenfeld that drive glaucoma or cataract.

These abnormalities are rare and often associated with extra-ocular malformations. Thus, a delay acquisitions may be present, secondary to sensory impairment, or directly related to a brain damage during development, leading to intellectual disability. The visual consequences of these malformations, as well as the frequency of extra-ocular and abnormalities of psychomotor development are still poorly known. Thus, predict the evolution the visual and neurological abilities of a child diagnosed with a congenital the eye will have been made during pregnancy or at birth and propose to these children a protocol well-defined care is proving very difficult at the moment. The aim of this study is to improve knowledge of these diseases by describing the course of visual and neuro-developmental functions.

The study should also:

1. Identify prognostic factors for the visual and neurological evolution of these diseases
2. Assess the impact of these eye defects on the quality of life of patients and their family
3. Search for correlations between the presence of certain genetic mutations and the appearanceocular or neuro-developmental abnormalities.

All these observations should improve the management of these diseases.

The patients involved are children and adults with congenital eye defects.

This will be a retrospective and prospective observational study. Any patient responding to criteria for inclusion and not satisfying the criteria for exclusion, duly informed and having given its consent, may be included in the study by his doctor.

ELIGIBILITY:
Inclusion Criteria:

* Newborns and/or children from birth to 7 years old, Children from 8 years old affected with the following ocular defects: anophthalmia, microphthalmia, aniridia or anterior segment dysgnesis.whose parents will have properly evaluated risks and benefits of the study and will be given an informed consent to participate the protocol.
* Patients affiliated to the "Régime National d'Assurance Maladie". Inclusion of foreign patients will be possible through the French inclusion centers when they agreed to be charged for all medical fees.
* Adults affected with the following ocular defects: anophthalmia, microphthalmia, aniridia or anterior segment dysgenesis
* Adult patients under guardianship whose guardians will have properly evaluated risks and benefits of the study and will be given an informed consent to participate the protocol. Indeed, intellectual disability may be associated with the ocular defects and we will need to include these patients in order to evaluate incidence of this event.
* Adult patients able to properly evaluate risks and benefits of the study and to give their informed consent to participate to the protocol.
* Adult parents of an affected child participating to the study and willing to participate to the inheritance study (results of DNA analysis).
* Inclusion of foreign patients will be possible through the French inclusion centres when they agreed to be charged for all medical fees.

Pregnant women can be included in the study

Exclusion Criteria:

* No exclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients from 0 to 7 years old We aim to include most patients born with a developmental ocular defect. Even if most ocular defects are diagnosed during the first months of age, patients could be included in the cohort until 7 years old.
  Patients over 8 years old: Affected adults and children over 8 years old will not be included in the follow-up subgroup.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2017-07-11 (Actual); Primary Completion 2037-07 (Estimated); Study Completion 2037-07 (Estimated)

PRIMARY OUTCOMES:
Visual acuity including distance and near vision, completed if necessary by a low vision evaluation with ETDRS scale, will be conducted with refraction under cycloplegia. | Up to 3 visits for patients < 6 years / Up to 2 visits for patients ≥ 6 years and < 8 years / 1 visit for patiens ≥ 8 years
An accurate description of the binocular vision by orthoptists | Up to 3 visits for patients < 6 years / Up to 2 visits for patients ≥ 6 years and < 8 years / 1 visit for patiens ≥ 8 years
Slit lamp examination and fundus with imaging will be useful to specify the disease. | Up to 3 visits for patients < 6 years / Up to 2 visits for patients ≥ 6 years and < 8 years / 1 visit for patiens ≥ 8 years
An ultrasound measurement will evaluate axial length of eyeball. | Up to 3 visits for patients < 6 years / Up to 2 visits for patients ≥ 6 years and < 8 years / 1 visit for patiens ≥ 8 years
Some imaging ocular techniques as videotopography (Pentacam) | Up to 3 visits for patients < 6 years / Up to 2 visits for patients ≥ 6 years and < 8 years / 1 visit for patiens ≥ 8 years
Some imaging ocular techniques as ultrabiomicroscopy to evaluate anterior segment | Up to 3 visits for patients < 6 years / Up to 2 visits for patients ≥ 6 years and < 8 years / 1 visit for patiens ≥ 8 years
Some imaging ocular techniques as macular OCT (spectral-domain optical coherence tomography) | Up to 3 visits for patients < 6 years / Up to 2 visits for patients ≥ 6 years and < 8 years / 1 visit for patiens ≥ 8 years
Imaging techniques to evaluate retina and optic nerve will be completed as appropriate due to the condition of the patient (low vision, nystagmus…). | Up to 3 visits for patients < 6 years / Up to 2 visits for patients ≥ 6 years and < 8 years / 1 visit for patiens ≥ 8 years
Neurological examination will be based on standard procedures (WISC at age 6 and WISCIV at age 10) | Up to 3 visits for patients < 6 years / Up to 2 visits for patients ≥ 6 years and < 8 years / 1 visit for patiens ≥ 8 years
Procedures adapted to visually impaired children when necessary | Up to 3 visits for patients < 6 years / Up to 2 visits for patients ≥ 6 years and < 8 years / 1 visit for patiens ≥ 8 years

SECONDARY OUTCOMES:
Ocular defects, unilateral or bilateral involvement | Up to 3 visits for patients < 6 years / Up to 2 visits for patients ≥ 6 years and < 8 years / 1 visit for patiens ≥ 8 years
Extraocular malformations | Up to 3 visits for patients < 6 years / Up to 2 visits for patients ≥ 6 years and < 8 years / 1 visit for patiens ≥ 8 years
Quality of life questionnaires | Up to 3 visits for patients < 6 years / Up to 2 visits for patients ≥ 6 years and < 8 years / 1 visit for patiens ≥ 8 years
  Short-Form Health Survey (SF-36) or equivalent adapted for children (SF-10)

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas NC CHASSAING, Dr, Principal Investigator — Centre de référence des maladies ophtalmologiques rares
Locations (1):
- RaDiCo-ACOEIL, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: Undecided